CLINICAL TRIAL: NCT05010057
Title: The Effect of New Zealand Blackcurrant (NZBC) Supplementation on Indices of Muscle Damage Following Strenuous Exercise
Brief Title: The Effect of New Zealand Blackcurrant (NZBC) Supplementation on Recovery Following Strenuous Exercise
Acronym: CurraNZ_MD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UEC/2015/112/FHMS
Record Dates: First submitted 2021-08-06; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Muscle Damage
Keywords: Exercise-induced muscle damage; Recovery; Supplementation; Oxidative stress; Anthocyanin; New Zealand blackcurrant

STUDY DESIGN:
Intervention Model Description: Randomised, parallel design.
Who Masked: Participant, Investigator
Masking Description: Coded, capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Zealand blackcurrants (NZBC) (Experimental): 1 NZBC capsule (containing 300 mg active cassis containing 105 mg of anthocyanins, i.e. 35-50 % delphinidin-3-rutinoside, 5-20 % delphinidin-3-glucoside, 30-45 % cyanidin-3-rutinoside, 3-10 % cyanidin-3-glucoside), consumed in the morning, for 12 days.
  Interventions: Dietary Supplement: New Zealand blackcurrants (NZBC)
- Placebo (PLA) (Placebo Comparator): 1 placebo capsule (containing 300 mg microcrystalline cellulose M102), consumed in the morning, for 12 days.
  Interventions: Dietary Supplement: Placebo (PLA)

INTERVENTIONS:
Dietary Supplement: New Zealand blackcurrants (NZBC) — NZBC capsules containing anthocyanin-rich blackcurrant extract
  Other Names: NZBC extract supplement (Health Currancy Ltd [UK] / CurraNZ Ltd [NZ])
  Arms: New Zealand blackcurrants (NZBC)
Dietary Supplement: Placebo (PLA) — Placebo capsules containing microcrystalline cellulose
  Other Names: Placebo capsules
  Arms: Placebo (PLA)

SUMMARY:
The study aims to examine the effect of a New Zealand blackcurrant (NZBC) supplement on markers of muscle damage and recovery following strenuous resistance exercise. The investigation will compare responses between an experimental (NZBC capsule, 300 mg/day) and placebo (PLA capsule, 300 mg sugar) group. Participants will attend a screening session where they will consent to the study, complete a pre-activity medical questionnaire and have their height, weight and resting blood pressure measured. If the participants meet the inclusion criteria they will perform a familarisation session on the muscle strength assessment. Participants will be randomized to NZBC or placebo groups, and consume one capsule in the morning (between 6-10 am) for 12 days. This is a double-blinded study, which means that the participant and the study team will not know which group the participants are assigned to until the study is over. On day 8 participants will perform a strenuous bout of upper body resistance exercise on the isokinetic dynamometer (exercise device). Muscle strength and soreness, arm circumference, and elbow range of motion will be measured, and a fasted blood sample will be collected, before and 24, 48, 72 & 96 hours after the muscle fatigue protocol (on days 9, 10, 11 & 12). A marker of muscle damage (creatine kinase [CK] concentration) will be measured in the blood samples. Participants will also be asked to complete a 6-day dietary record, beginning on day 7 and ending on the final day of testing (day 12).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 18 - 45 years old
* BMI: 19 - 29.9 kg/m2
* Healthy: no active disease process that could interfere with endpoints measured as determined by medical history

Exclusion Criteria:

* Smoking and tobacco use
* Takes medication [excluding contraception]
* BMI ≥ 30 kg/m2
* Hypertensive (diastolic > 90 and/or systolic blood pressure > 140 mmHg)
* History of musculoskeletal upper limb injuries
* Performs regular resistance exercise (> 2 sessions per week)
* Uses dietary supplements that could influence muscle recovery or function (e.g. protein supplements, antioxidants etc)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in creatine kinase (CK) concentration at 72 hours post-exercise | At baseline (pre-exercise) and 72 hours post-exercise.
  Serum biomarker for muscle damage
Change from baseline in creatine kinase (CK) concentration at 96 hours post-exercise | At baseline (pre-exercise) and 96 hours post-exercise..
  Serum biomarker for muscle damage

SECONDARY OUTCOMES:
Change in maximum voluntary contraction (MVC) from baseline to 96 hours post-exercise | At baseline (pre-exercise) and post-exercise time points (at 0, 24, 48, 72 and 96 hours respectively).
  Muscle function measure; maximal voluntary isometric contraction (torque, Nm) performed on isokinetic dynamometer
Change in rating of Delayed Onset of Muscle Soreness (DOMS) from baseline to 96 hours post-exercise | At baseline (pre-exercise) and post-exercise time points (at 24, 48, 72 and 96 hours respectively).
  Self-reported perception of muscle soreness using a visual analogue scale (VAS), from 'no soreness' [0 mm] on the left anchor point to 'extremely sore' [100 mm] on the right
Change in joint range of motion (ROM) from baseline to 96 hours post-exercise | At baseline (pre-exercise) and post-exercise time points (at 24, 48, 72 and 96 hours respectively).
  Elbow ROM measured using a goniometer
Change in mid arm circumference (MAC) from baseline to 96 hours post-exercise | At baseline (pre-exercise) and post-exercise time points (at 24, 48, 72 and 96 hours respectively).
  Mid-upper arm circumference measured at the midpoint of the distance from the acromion process (acromiale) to the olecranon process (radiale).

CONTACTS AND LOCATIONS:
Overall Officials: Julie EA Hunt, PhD, Principal Investigator — University of Surrey
Locations (1):
- Surrey Human Performance Institute, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will provide basic data spreadsheet upon request.